CLINICAL TRIAL: NCT00107237
Title: A Phase IB/II Multicenter, Two-Arm, Dose-Escalation Study of Oral AEE788 Administered in Combination With Oral RAD001 on a Continuous Once Daily Dosing Schedule in Adult Patients With First or Second Recurrent or Relapsing Glioblastoma Multiforme
Brief Title: AEE788 and Everolimus in Treating Patients With Recurrent or Relapsed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEE788A2106; UCLA-0409004-01; CDR0000422335 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — AEE 788; Everolimus

ARMS (2):
- AEE788 200 mg + RAD001 5 mg (Experimental): AEE788 200 mg qd, RAD001 5 mg qd
  Interventions: Drug: AEE788; Drug: everolimus
- AEE788 150 mg + RAD001 5mg (Experimental): AEE788 150 mg qd, RAD001 5 mg qod
  Interventions: Drug: AEE788; Drug: everolimus

INTERVENTIONS:
Drug: AEE788 — AEE788 was available in the form of a hard gelatin capsule of 50 mg or 100 mg strengths and packaged in bottles.
Drug: everolimus — Everolimus was formulated as tablets of 2.5 mg and 5 mg strength and supplied in blister packs.
  Other Names: RAD001

SUMMARY:
RATIONALE: AEE788 and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving AEE788 together with everolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of AEE788 when given together with everolimus and to see how well they work in treating patients with recurrent or relapsed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of AEE788 when administered in combination with 1 of 2 different doses of everolimus in patients with recurrent or relapsed glioblastoma multiforme.

Secondary

* Determine the safety and tolerability of this regimen, including acute and chronic toxic effects, in these patients.
* Determine the single-dose and repeated-dose pharmacokinetic profile of this regimen in these patients.
* Determine, preliminarily, the efficacy of this regimen, in terms of response rate, progression-free survival, and overall survival, in these patients. (Phase II)
* Determine the antiangiogenic effects of this regimen in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of AEE788.

* Phase I: Patients are assigned to 1 of 2 treatment groups.

  * Group 1: Patients receive oral AEE788 once daily and oral everolimus once daily on days 1-28.
  * Group 2: Beginning at the first occurrence of dose-limiting toxicity in group 1, patients receive AEE788 as in group 1 and a higher-dose of oral everolimus once daily on days 1-28.

In both groups, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients per group receive escalating doses of AEE788 until the maximum tolerated dose is determined.

* Phase II: Patients are assigned to 1 of 2 treatment groups according to eligibility for surgery.

  * Group 1 (eligible for tumor biopsy, surgical resection, or tumor debulking): Patients receive oral AEE788 once daily at the MTD and oral everolimus once daily for 5-9 days. Patients then undergo surgery. Beginning 15-21 days after surgery, patients receive oral AEE788 and oral everolimus once daily on days 1-28.
  * Group 2 (ineligible for surgery): Patients receive oral AEE788 once daily at the MTD and oral everolimus once daily on days 1-28.

In both groups, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. In both phases, if treatment with AEE788 or everolimus is stopped due to toxicity, patients may continue to receive AEE788 or everolimus alone once daily.

After the completion of study treatment, patients are followed every 3 months for as long as the investigator deems necessary.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme, meeting 1 of the following criteria:

  * Phase I

    * In first or second recurrence or relapse
    * At least 1 measurable or evaluable enhancing lesion by gadolinium MRI (Gd-MRI) of the brain within the past 3 weeks
  * Phase II, group 1

    * In first or second recurrence or relapse by Gd-MRI of the brain within the past 3 weeks
    * Requires tumor biopsy OR surgical resection for tumor debulking or for confirmation of recurrence
  * Phase II, group 2

    * In first recurrence or relapse
    * At least 1 bidimensionally measurable enhancing lesion (≥ 1.5 cm^2 using product of the largest perpendicular diameters) by Gd-MRI of the brain within the past 3 weeks
* Multifocal disease allowed

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* No acute or chronic liver disease

Renal

* Total calcium (corrected) normal*
* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min
* No proteinuria by dipstick OR
* Total urinary protein ≤ 500 mg AND creatinine clearance ≥ 50 mL/min by 24-hour urine collection
* No acute or chronic renal disease NOTE: *Supplements allowed

Cardiovascular

* LVEF ≥ 45% by MUGA or echocardiogram
* No complete left bundle branch block
* No requirement for a cardiac pacemaker
* No congenital long QT syndrome
* No ventricular or atrial tachyarrhythmias
* No clinically significant resting bradycardia, defined as < 50 beats per minute
* QTc ≤ 480 msec by ECG
* No right bundle branch block and left anterior hemiblock (bifascicular block)
* No uncontrolled hypertension OR history of labile hypertension
* No unstable angina pectoris OR angina pectoris occurrence within the past 3 months
* No congestive heart failure
* No acute myocardial infarction within the past 3 months
* No history of poor compliance with an antihypertensive regimen
* No other impaired cardiac function or clinically significant cardiac disease

Gastrointestinal

* No unresolved diarrhea ≥ grade 2
* No impairment of gastrointestinal (GI) function or GI disease that would significantly alter absorption of study drugs, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea
  * Vomiting
  * Malabsorption syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* Potassium normal*
* Magnesium normal*
* Phosphorus normal*
* Cholesterol ≤ 300 mg/dL (treatment allowed)
* Triglycerides ≤ 2.5 times ULN (treatment allowed)
* No known HIV positivity
* No peripheral neuropathy ≥ grade 2
* No uncontrolled diabetes
* No active or uncontrolled infection
* No other severe and/or uncontrolled medical condition that would preclude study participation or compliance
* No contraindication to MRI, including any of the following:

  * Cardiac pacemaker
  * Ferromagnetic metal implants other than those approved as safe for use with magnetic resonance scanners (e.g., some types of aneurysm clips or shrapnel)
  * Claustrophobia
  * Obesity exceeding magnetic resonance equipment limits
* No other clinically significant primary malignancy requiring active intervention NOTE: *Supplements allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior hematopoietic colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) except epoetin alfa
* More than 2 weeks since prior immunotherapy and recovered
* No concurrent biologic therapy
* No concurrent prophylactic hematopoietic growth factors (e.g., G-CSF or GM-CSF) unless approved by the study sponsor

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior polifeprosan 20 with carmustine implant (Gliadel® wafer) allowed
* No other concurrent chemotherapy

Endocrine therapy

* Must be on stable or deceasing doses of steroids for at least 7 days before baseline Gd-MRI of the brain and before starting study drug
* No concurrent tamoxifen

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* More than 1 week since prior tumor biopsy
* More than 2 weeks since prior surgical resection
* More than 2 weeks since prior major non-CNS surgery and recovered
* No prior small bowel resection

Other

* At least 2 weeks since prior and no concurrent enzyme-inducing anticonvulsant drugs
* More than 4 weeks since prior investigational drugs and recovered
* No prior epidermal growth factor receptor- or ErbB-2-directed therapy (phase II only)
* No prior vascular endothelial growth factor (VEGF) or VEGF receptor-directed therapy (phase II only)
* No prior mTOR-directed therapy (phase II only)
* No concurrent therapeutic warfarin
* No concurrent treatment with any medication that may prolong QT interval, including any of the following:

  * Quinidine
  * Procainamide
  * Disopyramide
  * Amiodarone
  * Sotalol
  * Bretylium
  * Ibutilide
  * Thioridazine
  * Mesoridazine
  * Chlorpromazine
  * Amitriptyline
  * Imipramine
  * Desipramine
  * Doxepin
  * Erythromycin
  * Clarithromycin
  * Ketoconazole
  * Halofantrine
  * Quinine
  * Chloroquine
  * Mefloquine
  * Moxifloxacin
  * Gatifloxacin
  * Pimozide
  * Risperidone
  * Ziprasidone
  * Venlafaxine
  * Maprotiline
  * Lithium
  * Pentamidine
  * Droperidol
  * Dolasetron
* No concurrent digoxin or verapamil
* No concurrent tacrolimus
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of AEE788

SECONDARY OUTCOMES:
Safety
Tolerability
Single-dose and repeated-dose pharmacokinetic profile
Efficacy (response rate, progression-free survival, and overall survival)
Antiangiogenic effects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Duke Univaersity Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center/University of Texas, Houston, Texas